CLINICAL TRIAL: NCT06707896
Title: Phase I, Open-Label Study of Autologous Mutant KRAS-redirected T-cell Receptor Cells (TCR1020-CD8)
Brief Title: TCR1020-CD8 T Cells in KRAS-mutated Cancers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative decision
Sponsor: University of Pennsylvania (Other)
Collaborators: Stand Up To Cancer (Other); Lustgarten Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18224
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 (Experimental): After lymphodepleting chemotheerapy subjects will recieve a dose of 3 x 10(8) TCR1020-CD8 T cells
  Interventions: Drug: TCR1020-CD8 T cells
- Dose Level -1 (Experimental): After lymphodepleting chemotheerapy subjects will recieve a dose 1 x 10(8) TCR1020-CD8 T cells
  Interventions: Drug: TCR1020-CD8 T cells
- Dose Level 2 (Experimental): After lymphodepleting chemotheerapy subjects will recieve a dose 1 x 10(9) TCR1020-CD8 T cells
  Interventions: Drug: TCR1020-CD8 T cells
- Dose Level 3 (Experimental): After lymphodepleting chemotheerapy subjects will recieve a dose 3 x 10(9) TCR1020-CD8 T cells
  Interventions: Drug: TCR1020-CD8 T cells

INTERVENTIONS:
Drug: TCR1020-CD8 T cells — TCR1020-CD8 T cells are autologous mKRAS-redirected CD8+ T cells engineered using a lentiviral vector to express a TCR with specificity for HLA-restricted mKRAS G12V epitopes restricted to the HLA-A*11:01 molecule.

SUMMARY:
This is a Phase I, open-label dose finding study to assess the safety, manufacturing feasibility, and preliminary efficacy of TCR1020-CD8 T cells in patients with KRAS-mutated cancers. Initially, patients with KRAS G12V mutation positive metastatic pancreatic adenocarcinoma or colorectal cancer will be targeted for participation. Up to 4 total dose levels will be evaluated using a 3+3 dose escalation design.

DETAILED DESCRIPTION:
This is a Phase I, open-label dose finding study to assess the safety, manufacturing feasibility, and preliminary efficacy of TCR1020-CD8 T cells in patients with KRAS-mutated cancers.

Initially, patients with KRAS G12V mutation positive metastatic pancreatic adenocarcinoma or colorectal cancer will be targeted for participation. Up to 4 total dose levels will be evaluated using a 3+3 dose escalation design as described in protocol Section 3.1.

In order to allow for appropriate monitoring/assessment of toxicities, the TCR1020-CD8 T cell infusions will be staggered as follows:

* The TCR1020-CD8 T cell infusions for the first two subjects treated at each dose level must be staggered by at least 28 days.
* If there are no emergent safety concerns identified in the first subject treated at each dose level, infusions of the 2ⁿᵈ and 3ʳᵈ subjects at that dose level may occur in parallel.
* A stagger will occur after every 3ʳᵈ subject is infused to allow for formal DLT assessments to be performed and the dose level assignment for the next subject to be confirmed.
* In the event 1 DLT is identified at a dose level (e.g., 1 DLT/3 evaluable subjects), formal DLT evaluations must be completed after each additional TCR1020-CD8 T cell infusion to evaluate potential dose de-escalation rules. As such, subsequent TCR1020-CD8 T cell infusions within that same dose level must be staggered by a minimum of 28 days.
* If emergent safety concerns are identified, an ad hoc DLT evaluation may be triggered at the request of the Safety Review Committee (SRC). The purpose, scope and composition of the SRC is further defined in protocol Section 3.3.

The DLT observation period is 28 days post-TCR1020-CD8 T cell infusion (Day 0). Formal DLT evaluations will be performed after the 3ʳᵈ DLT-evaluable subject at each dose level completes this 28-day DLT monitoring window. These assessments will be performed by the Safety Review Committee (SRC), comprised of the Clinical PI and Sponsor Medical Director, in accordance with the definitions/requirements in protocol Section 8.1.6. The SRC will trigger a decision regarding dose level advancement, expansion, or dose de-escalation. The highest dose at which 0 or 1 DLT occurs in 6 DLT-evaluable subjects will be declared the maximum tolerated dose (MTD).

Subjects must receive the dose of TCR1020-CD8 T cells as per their dose level assignment in order to be considered DLT-evaluable for dose escalation decisions and MTD determination. Subjects who do not receive the dose of TCR1020-CD8 T cells as per their dose level assignment will not be considered DLT-evaluable for this purpose and will be replaced at that dose level. However, these subjects will still be followed per protocol and included in the overall safety analysis, as wellas the analyses of secondary and exploratory endpoints.

Retreatment Infusions:

The Retreatment Phase will remain closed until sufficient safety data is available in initial subjects, and DSMB and FDA approval to open Retreatment has been received.

Subjects who have demonstrated clinical benefit after their initial TCR1020-CD8 T cell infusion(e.g., minimum disease response of stable disease, etc.) may also be eligible to receiveretreatment with TCR1020-CD8 cells at the physician-investigator's discretion. The TCR1020-CD8retreatment dose administered must either be a). the T cell dose that the subject previouslyreceived without DLTs, or b). a T cell dose that is less than or equal to a dose level that has beenevaluated for safety in ≥ 3 other subjects without evidence of DLTs. As retreatment infusions willnot be used for formal DLT assessments/MTD determination, there are no protocol-definedstaggering requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age
2. Patients with one of the following diagnoses:

   1. Histologically confirmed metastatic pancreatic adenocarcinoma
   2. Histologically confirmed metastatic colorectal cancer
3. HLA-A*11:01 positive
4. KRAS G12V mutation positive disease as confirmed by a CLIA certified laboratory.
5. Received prior treatment for their primary malignancy as follows:

   1. Pancreatic Cancer Patients: At least one prior line of standard of care therapy for advanced stage disease
   2. Colorectal Cancer Patients: At least two prior lines of standard of care therapy for advanced stage disease.
6. Evidence of active disease within 8 weeks of physician-investigator confirmation of eligibility.
7. Adequate organ function within 4 weeks of eligibility confirmation by a physician-investigator defined as:

   1. Serum creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 50 cc/min per the Cockcroft-Gault Equation; Patient must not be on dialysis.
   2. ALT/AST ≤ 5 x ULN (patients with liver metastases) or ALT/AST ≤ 2.5 x ULN (patients without liver metastases)
   3. Direct bilirubin ≤ 2 mg/dL, unless the subject has Gilbert's syndrome (if so, direct bilirubin must be ≤3.0 mg/dL)
   4. Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO
   5. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air
8. Patients must have adequate hematologic reserve within 4 weeks of eligibility confirmation by a physician-investigator and must not be dependent on transfusions to maintain these hematologic parameters. Adequate hematologic reserve is defined as:

   1. Hemoglobin ≥ 8 g/dL
   2. Absolute neutrophil count ≥ 1000/μL
   3. Platelet count ≥ 75,000/μL
9. ECOG Performance Status that is either 0 or 1.
10. Signed, written informed consent
11. Participants of reproductive potential must agree to use acceptable birth control methods, asdescribed in protocol Section 4.3.

Exclusion Criteria:

1. Active hepatitis B or hepatitis C infection
2. Any other active, uncontrolled infection.
3. Class III/IV cardiovascular disability according to the New York Heart Association Classification (see Appendix 5 of the protocol for full details).
4. Severe, active co-morbidity that in the opinion of the physician-investigator would preclude participation in the study.
5. Active invasive cancer, other than the proposed cancer included in the study, within 2 years prior to eligibility confirmation by a physician-investigator. [Note: non-invasive cancers treated with curative intent (e.g., non-melanoma skin cancer) may still be eligible].
6. Pregnant or nursing (lactating) patients. Participants of reproductive potential must agree to use acceptable birth control methods, as described in protocol Section 4.3.
7. Patients requiring chronic treatment with systemic steroids or immunosuppressant medications. Low-dose physiologic replacement therapy with corticosteroids equivalent to prednisone 10 mg/day or lower, topical steroids and inhaled steroids are acceptable. For additional details regarding use of steroid and immunosuppressant medications, please see protocol Section 5.6.
8. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10mg of prednisone. Patients with autoimmune neurologic diseases (such as MS) will be excluded.
9. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2044-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with dose limiting toxicities (DLTs) | 28 days after TCR1020-CD8 T cells
Determination of maximum tolerated does (MTD) | 28 days after TCR1020-CD8 T cells
Incidence of Adverse Events as assessed by CTCAE v5.0 | Up to 15 years

SECONDARY OUTCOMES:
Percentage of manufacturing products that meet release criteria | Up to 3 years
Overall Response Rate (ORR) | Up to one year
Duration of Response (DOR) | Up to one year
Progression Free Survival (PFS) | Up to 15 years
Overall Survival (OS) | Up to 15 years